CLINICAL TRIAL: NCT00144573
Title: An Open-Label, Clinical Pharmacology Study to Evaluate the Safety and PK of MRA in Patients With RA With Renal Impairment
Brief Title: Clinical Pharmacology Study of MRA in Patient With Rheumatoid Arthritis (RA) With Renal Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA221JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

INTERVENTIONS:
Drug: MRA(Tocilizumab)

SUMMARY:
This is an open-label, clinical pharmacology study to evaluate the safety and PK of MRA in patients with RA with Renal Impairment.

ELIGIBILITY:
Inclusion criteria

* Patients who are diagnosed with RA according to the 1987 ACR (American College of Rheumatology) classification criteria
* Patients with RA at least 6 months prior to enrollment
* Patients with a creatinine clearance not less than 10 mL/min but no higher than 80 mL/min

Exclusion criteria

* Patients with Class IV Steinbrocker functional impairment at enrollment
* Patients who are undergoing dialysis
* Patients who have been treated for the underlying disease with a biological agent, such as infliximab or etanercept, and have been receiving treatment with leflunomide, within 12 weeks before treatment with the investigational product

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-01; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
20% improvement based on the ACR criteria compared with the baseline value. | throughout study

SECONDARY OUTCOMES:
Time courses taken from baseline values for DAS28, for ACR20%, 50%, and 70% improvement, and for each ACR core set variable. | Week 0, Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical